CLINICAL TRIAL: NCT04420533
Title: Comparative Study Between Behavior Therapy and Behavior Therapy Plus Mirabegron 50mg in Sexually Active Men With Bothersome Overactive Bladder Symptoms - A Multicenter, Randomized Study
Brief Title: Comparative Study Between Behavior Therapy and Behavior Therapy Plus Mirabegron in Sexually Active Men With OAB Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202000790A3
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Urinary Bladder, Overactive; Sexual Behavior; Sexual Activity; Behavior Therapy; Sexual Function Disturbances
Keywords: overactive bladder; mirabegron 50mg
MeSH Terms: conditions — Urinary Bladder, Overactive; Sexual Behavior; Sexual Dysfunctions, Psychological | interventions — Behavior Therapy; mirabegron

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-center, randomized, open label study in sexually active male OAB patients treated with behavior therapy alone or behavior therapy plus mirabegron 50mg OD in a 1:2 ratio.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavior therapy alone (Active Comparator): Behavior therapy alone
  Interventions: Behavioral: Behavior therapy alone
- Behavior therapy plus mirabegron 50mg (Experimental): Behavior therapy plus Betmiga prolonged-release tablets (mirabegron) 50mg QDAC PO
  Interventions: Behavioral: Behavior therapy alone; Drug: Mirabegron 50 MG Extended Release Oral Tablet

INTERVENTIONS:
Behavioral: Behavior therapy alone — 1. reduction of fluid intake at specific times aimed at reducing urinary frequency when most inconvenient;
  2. moderation of intake of caffeine or alcohol, which may have a diuretic and irritant effect, thereby increasing fluid output and enhancing frequency, urgency and nocturia;
  3. use of relaxed and double-voiding techniques;
  4. urethral milking to prevent post-micturition dribble;
  5. distraction techniques such as penile squeeze, breathing exercises, perineal pressure, and mental tricks to take the mind off the bladder and toilet, to help control storage symptoms;
  6. bladder retraining that encourages men to hold on when they have sensory urgency;
  7. reviewing the medication and optimising the time of administration or substituting drugs for others that have fewer urinary effects (these recommendations apply especially to diuretics);
  8. providing necessary assistance when there is impairment of dexterity, mobility or mental state;
  9. treatment of constipation.
Drug: Mirabegron 50 MG Extended Release Oral Tablet — Betmiga prolonged-release tablets (mirabegron) 50mg QDAC PO
  Other Names: Mirabegron 50 MG
  Arms: Behavior therapy plus mirabegron 50mg

SUMMARY:
The objective of this study is to evaluate and compare the therapeutic effects on OAB symptoms, and sexual functions, in terms of erectile function and ejaculatory function, in sexually active OAB male treated with behavior therapy or behavior therapy plus Mirabegron (50 mg).

DETAILED DESCRIPTION:
Overactive bladder (OAB) syndrome is a subset of storage-predominant lower urinary tract symptoms (LUTS) and has a significant impact on quality of life. Men with OAB generally experience a reduced quality of life, which may include a negative impact on sexual function. A previous study revealed that OAB is associated with erectile dysfunction (ED; prevalence odds ratio, 1.5; 95% confidence interval, 1.1-2.2) to a level comparable with that of hypertension or diabetes, both of which are known risk factors for ED. Furthermore, men with OAB were nine and seven times more likely to report diminished sexual enjoyment and decreased sexual activity, respectively, due to urinary symptoms than men without urinary symptoms.

Behavior therapies are designed as first- line treatment for the treatment of OAB with or without concomitant medication. Mirabegron, a selective β3 adrenoceptor agonist, is indicated for the treatment of OAB. Earlier research studying the role and distribution of β3-adrenoreceptors revealed that the receptors exert other physiological functions such as lipolysis and are present not only in adipose tissue but also in human gall bladder, colon, prostate, skeletal muscles and corpus cavernosum (CC) smooth muscles. It was found that activation by a selective experimental β3-receptor agonist, BRL 37344, elicited relaxation of human CC smooth muscle via a cGMP-dependent but NO-independent mechanism, leading to observable β3-receptor-mediated vasorelaxant tone of CC. The potential effect of β3-receptor agonism at human CC mediated by highly selective mirabegron in both human CC and rat CC that mirabegron markedly relaxed isolated CC strips by activating β3-adrenoceptors localized in cavernosal smooth muscle cells, independently of the NO-cGMP pathway. Recently, intra-cavernosal injection of mirabegron improved erectile function and neurogenic relaxation of corpus cavernosum in diabetic rats.

These early results have spurred research interest in mirabegron-induced CC relaxation and encouraged further clinical studies observing and evaluating the effect of mirabegron on male sexual function. Researchers at Johns Hopkins University has recently completed recruitment of a phase 1 interventional trial (NCT02916693) that aimed to address the hypothesis that activation of β3-adrenoceptors by mirabegron offers an alternative pharmacologic pathway for the treatment of erectile dysfunction. A preliminary small-scale prospective interventional study including 128 male LUTS patients treated with mirabegron 50 mg, 34 of whom had diagnosis of OAB and were sexually active, showed that mirabegron usage did not improve erectile function, as evaluated by International Index of Erectile Function (IIEF-5 4.9% decrease at 4-week; p = 0.106, and 9.1% decrease at 12-week follow-up; p = 0.077). However, the IIEF-5 was significantly decreased in the higher baseline IIEF-5 (≥17) group (11.7% decrease; p = 0.044), noncoronary artery disease (13.2%; p = 0.007) group and non-DM group (13.9% decrease; p = 0.021) at 12-week follow-up.

The accumulated research output warrants the initiation of a prospective study involving a larger patient cohort to evaluate the effect of mirabegron on male sexual function in addition to alleviate OAB symptoms. The objective of this study is to evaluate and compare the therapeutic effects on OAB symptoms, and sexual functions, in terms of erectile function and ejaculatory function, in sexually active OAB male treated with behavior therapy or behavior therapy plus Mirabegron (50 mg).

ELIGIBILITY:
Inclusion Criteria:

* Sexually active men with OAB ≥ 20 years
* Diagnosed with OAB based on OABSS (OABSS urgency score of ≥2 and sum score of ≥3)
* Patients can sign informed consent and record voiding diary

Exclusion Criteria:

* Concurrent use of PDE5 inhibitor or testosterone therapy during study period
* History of stress urinary incontinence
* Neurologic conditions associated with OAB symptoms
* Evidence of active urinary tract infection or urinary tract stone at screening
* Confirmed or suspected genitourinary tract or pelvic malignancy
* Genitourinary tract operation during the 3-month period prior to baseline
* Postvoid residual urine volume (PVR) ≥ 100 mL
* History of uncontrolled hypertension (systolic >180 mmHg and/or diastolic >110 mmHg)
* History of intolerance to mirabegron
* History of medical conditions or presence of patient factors that, in the judgement of the investigator, would preclude adherence to study protocol
* Patient had received intravesical onabotulinumoxinA treatment within recent 6 months

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in OABSS at Week 12 | Baseline and Week 12
  Change from baseline in OABSS (Overactive Bladder Symptom Score) at Week 12 (lower OABSS score represent a better outcome)
Change from baseline in IIEF-5 at Week 12 | Baseline and Week 12
  Change from baseline in IIEF-5 (International Index of Erectile Function) at Week 12 (higher IIEF-5 score represent a better outcome)

SECONDARY OUTCOMES:
Change from baseline in OABSS at Week 4 | Baseline and Week 4
  Change from baseline in OABSS (Overactive Bladder Symptom Score) at Week 12 (lower OABSS score represent a better outcome)
Change from baseline in IIEF-5 at Week 4 | Baseline and Week 4
  Change from baseline in IIEF-5 (International Index of Erectile Function) at Week 12 (higher IIEF-5 score represent a better outcome)
Change from baseline in MSHQ-EjD Short Form score at Week 4 | Baseline and Week 4
  Change from baseline in MSHQ-EjD (Male Sexual Health Questionnaire -Ejaculatory Domain) Short Form score at Week 4 (higher MSHQ-EjD Short Form Q1-Q3 sum scores represent a better outcome; lowerer MSHQ-EjD Short Form Q4 score represent a better outcome)
Change from baseline in MSHQ-EjD Short Form score at Week 12 | Baseline and Week 12
  Change from baseline in MSHQ-EjD (Male Sexual Health Questionnaire -Ejaculatory Domain) Short Form score at Week 12 (higher MSHQ-EjD Short Form Q1-Q3 sum scores represent a better outcome; lower MSHQ-EjD Short Form Q4 score represent a better outcome)
Net change of Frequency episode, nocturia episode, urgency episode, UUI episodes in 3-day voiding diary from baseline to 1 and 3 months after the treatment day | Baseline, Week 4 and Week 12
  Net change of Frequency episode, nocturia episode, urgency episode, UUI episodes in 3-day voiding diary from baseline to 1 and 3 months after the treatment day (lower episode represent a better outcome)
Net change of Qmax from baseline to 1 and 3 months after the treatment day | Baseline, Week 4 and Week 12
  Net change of maximum flow rate (Qmax) from baseline to 1 and 3 months after the treatment day (higher Qmax and voided volume represent a better outcome)
Net change of voided volume from baseline to 1 and 3 months after the treatment day | Baseline, Week 4 and Week 12
  Net change of voided volume from baseline to 1 and 3 months after the treatment day (higher voided volume represent a better outcome)
Net change of PVR volume from baseline to 1 and 3 months after the treatment day | Baseline, Week 4 and Week 12
  Net change of postvoid residual (PVR) volume from baseline to 1 and 3 months after the treatment day (lower PVR represent a better outcome)
Net change of IPSS from baseline to 1 and 3 months after the treatment day | Baseline, Week 4 and Week 12
  Net change of IPSS (International prostate symptom score) from baseline to 1 and 3 months after the treatment day (lower IPSS represent a better outcome)
Net change of PPBC score from baseline to 1 and 3 months after the treatment day | Baseline, Week 4 and Week 12
  Net change of PPBC score (Patient perception of bladder condition) from baseline to 1 and 3 months after the treatment day (lower PPBC represent a better outcome)
Net changes of the GRA | Baseline, Week 4 and Week 12
  Global response assessment (GRA) of satisfaction by the patient (categorized into -3, -2, -1, 0, 1, 2, 3, indicating markedly worse to markedly improved) at 1 and 3 months after the treatment day. An improvement of GRA by 2 scales is considered effective.

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Tang Hsieh, MD, Study Chair — Institutional Review Board Chang Gung Medical Foundation
Locations (1):
- Chang Gung Memorial Hospital, Chang Gung University College of Medicine, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Chuang YC, Liu SP, Lee KS, Liao L, Wang J, Yoo TK, Chu R, Sumarsono B. Prevalence of overactive bladder in China, Taiwan and South Korea: Results from a cross-sectional, population-based study. Low Urin Tract Symptoms. 2019 Jan;11(1):48-55. doi: 10.1111/luts.12193. Epub 2017 Oct 2. PMID 28967230
- [Background] Irwin DE, Milsom I, Reilly K, Hunskaar S, Kopp Z, Herschorn S, Coyne KS, Kelleher CJ, Artibani W, Abrams P. Overactive bladder is associated with erectile dysfunction and reduced sexual quality of life in men. J Sex Med. 2008 Dec;5(12):2904-10. doi: 10.1111/j.1743-6109.2008.01000.x. PMID 19090944
- [Background] Coyne KS, Sexton CC, Thompson C, Kopp ZS, Milsom I, Kaplan SA. The impact of OAB on sexual health in men and women: results from EpiLUTS. J Sex Med. 2011 Jun;8(6):1603-15. doi: 10.1111/j.1743-6109.2011.02250.x. Epub 2011 Apr 14. PMID 21492396
- [Background] Yamaguchi O, Chapple CR. Beta3-adrenoceptors in urinary bladder. Neurourol Urodyn. 2007;26(6):752-6. doi: 10.1002/nau.20420. PMID 17600372
- [Background] Cirino G, Sorrentino R, di Villa Bianca Rd, Popolo A, Palmieri A, Imbimbo C, Fusco F, Longo N, Tajana G, Ignarro LJ, Mirone V. Involvement of beta 3-adrenergic receptor activation via cyclic GMP- but not NO-dependent mechanisms in human corpus cavernosum function. Proc Natl Acad Sci U S A. 2003 Apr 29;100(9):5531-6. doi: 10.1073/pnas.0931347100. Epub 2003 Apr 21. PMID 12707413
- [Background] Gur S, Peak T, Yafi FA, Kadowitz PJ, Sikka SC, Hellstrom WJ. Mirabegron causes relaxation of human and rat corpus cavernosum: could it be a potential therapy for erectile dysfunction? BJU Int. 2016 Sep;118(3):464-74. doi: 10.1111/bju.13515. Epub 2016 May 26. PMID 27124860
- [Background] Yilmaz-Oral D, Kaya-Sezginer E, Askin D, Hamurtekin Y, Gur S. Mirabegron, A Selective beta3-Adrenoceptor Agonist Causes an Improvement in Erectile Dysfunction in Diabetic Rats. Exp Clin Endocrinol Diabetes. 2021 Mar;129(4):296-302. doi: 10.1055/a-0869-7493. Epub 2019 Apr 12. PMID 30978726
- [Background] Wu TH, Shen YC, Lee WC, Wang HJ, Chuang YC. Effect of mirabegron on erectile function in sexually active men with bothersome overactive bladder symptoms. J Chin Med Assoc. 2020 Jan;83(1):55-59. doi: 10.1097/JCMA.0000000000000208. PMID 31567878
- See also: Management of Non-neurogenic Male LUTS. European Association of Urology, 2019 Guidelines — https://uroweb.org/guideline/treatment-of-non-neurogenic-male-luts/
- See also: ClinicalTrials.gov Identifier NCT02916693, Mirabegron For Erectile Dysfunction — https://clinicaltrials.gov/ct2/show/NCT02916693?term=NCT02916693&draw=2&rank=1

DOCUMENTS (2):
  • Study Protocol (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT04420533/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT04420533/SAP_001.pdf